CLINICAL TRIAL: NCT05571553
Title: E-health and People Living With Major Neurocognitive Disorder: A Study of the Effects of the CARE© and ESOGER© Applications
Brief Title: E-health and People Living With Major Neurocognitive Disorder - CARE© and ESOGER© Applications
Acronym: TNCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Senior researcher, Director of laboratory, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-1625
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Major Neurocognitive Disorder; Frailty
Keywords: E-Health
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Phase 1
  This is an experimental study of the randomized, longitudinal, prospective clinical trial type with a 3-month follow-up, open, in parallel groups (intervention versus control), carried out in people living with an MNCD and their family caregivers.
  Number of participants : 120
  Phase 2
  This is a randomized, longitudinal, prospective, clinical trial with a 6-month follow-up, open, in parallel groups (intervention versus control), carried out in people living with an MNCD.
  The total number of participants needed will be re-evaluated following analysis of the results obtained in Phase 1. We estimate at this time that a total of 40 participants per group, for a total of 80 people, is the number of participants needed for this study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Phase 1
  * Participants will assess their health status, at home, at recruitment (M0) and at 3 months (M3) with CARE© with the help of their family caregivers.
  * The principal investigator or a representative will contact them by phone within 5 days of the CARE© assessment to complete ESOGER.
  Phase 2
  * Participants will assess their health status, at home, at recruitment (M0), at 3 months (M3), and at 6 months (M6) on the CARE© application with the help of their family caregivers. An additional assessment will take place over the phone by the principal investigator or one of his representatives.
  * If their health status is considered fragile, then individuals will be contacted by phone by the PI or one of his representatives to complete the ESOGER© questionnaire (at M0, M3 and M6).
  Interventions: Other: Recommendations and reorientation towards healthcare resources
- Control group (No Intervention): Phase 1
  * Participants will assess their health status, by telephone, at recruitment (M0) and at 3 months (M3) with CARE© with the help of their family caregivers.
  * The principal investigator or a representative will contact them by phone within 5 days of the CARE© assessment to complete ESOGER.
  Phase 2
  * Participants will assess their health status, at home, at recruitment (M0), at 3 months (M3), and at 6 months (M6) on the CARE© application with the help of their family caregivers. An additional assessment will take place over the phone by the principal investigator or one of his representatives.
  * If their health status is considered fragile, then individuals will be contacted by phone by the PI or one of his representatives to complete the ESOGER© questionnaire (at M0, M3 and M6).

INTERVENTIONS:
Other: Recommendations and reorientation towards healthcare resources — Phase 1
  * After completing the CARE© questionnaire, participants will be given recommendations.
  * After the ESOGER© assessment, the participants will be contacted by the Red Cross who will set up the necessary interventions. They will be informed of the results of the assessments made.
  Phase 2
  * After completing the CARE© questionnaire, participants will be given recommendations.
  * If their health status is judged fragile by the CARE© score, and after the ESOGER© assessment, the participants will be contacted by the Red Cross who will set up the necessary interventions. They will be informed of the results of the assessments.
  For both phases, after 3 (6) months, the participants of the Control group will benefit from the recommendations following the CARE© assessment done at M3 (M6), and if necessary from the ESOGER© assessment and the Red Cross intervention. Throughout the study, they will continue to receive their conventional care.
  Arms: Intervention group

SUMMARY:
The care pathways of people living with major neurocognitive disorders (MNCD) are often inadequate due to poor access to resources, long delays, and resources that are poorly adapted to expectations and needs. This situation was exacerbated during the coronavirus disease (COVID-19) pandemic due to the reduction of available resources and care provider burnout. People living with MNCD are at risk of becoming more fragile, which can lead to emergency room visits and hospitalizations, and significantly alter the quality of life of the dyad (family caregiver and the person being cared for). Intervening earlier in the care pathway would make it possible to avoid the aggravation of pathologies associated with MNCD and hospitalizations.

The reorganization of activities imposed by the social distancing measures due to the pandemic has shown that e-health is a solution to maintain access to resources for people living with chronic conditions such as MNCD. We have been working since the beginning of the pandemic on the development of two complementary health applications for seniors and their dyads: the self-assessment questionnaire on frailty (CARE©) and the Evaluation et orientation SOcio-GÉRiatrique (ESOGER©) questionnaire :

* CARE© is made by the dyad, allowing to identify a state of frailty and the risks related to it. It relies on the active participation of the user and is deployed in the form of an application.
* ESOGER© is a standardized hetero-questionnaire filled out remotely, during a telephone call, by a community organization worker with the user and/or his/her caregiver. It is a tool for first contact, listening and accompanying a user, which makes it possible to determine whether the needs for care and services are being met, to prioritize the needs, to trigger the implementation of care and services, and to make the link with the organizations providing care and services.

The objectives of this study are to examine the effects of CARE© combined with ESOGER© on the state of physical and mental frailty, loss of autonomy, quality of life, and consumption of health services and care resources in people living with a major neurocognitive disorder (MNCD).

DETAILED DESCRIPTION:
This study includes two phases. The first phase is a feasibility study that aims to assess the behavior of users in relation to digital tools. Phase 2 will focus on evaluating the effects of the recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Be 65 years old or older.
* Have been previously diagnosed of MNCD (major neurocognitive disorder).
* Have a caregiver.
* Live in Montreal.
* Live at home or in a residence for seniors (RPA) in a non-medicalized area.
* Have an internet connection.
* Have a computer, or a touch pad or a smart phone.
* Understand French or English orally and in writing. The speakers are French and/or English speaking, and the questionnaires are only available in these 2 languages.

Exclusion Criteria:

* Participate in a concurrent investigational clinical study, to avoid interference with our study
* Live in a Residential and Long-Term Care Center (CHSDL) or in a medical sector in an RPA

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
CARE© Score | 8 months
  Measure of frailty via a standardized self-questionnaire consisting of 22 simple questions.
  The CARE© score ranges from 0 (no deficits) to 21 (maximum cumulative deficits). This score has been segmented into 3 levels according to a validated approach in order to determine 3 levels of frailty which are :
  * The robust level: score between 0 and 1.
  * The pre-fragile level: score between 2 and 4.
  * The fragile level: score > 5.
  For phase 1 : evaluated at M0 and M3, and the variation between M0 and M3. For phase 2 : evaluated at M0, M3 and M6, and the variation between the three periods.
Response Rate to CARE© questionnaires | 4 months
  Response Rate to CARE© questionnaires and the time required to complete the questionnaires.
  For phase 1 only.

SECONDARY OUTCOMES:
BGA Score | 8 months
  Measure of physical frailty using the Brief Geriatric Assessment (BGA) questionnaire with a score that ranges from 0 (no fragility) to 14 (severe fragility).
  For both phases.
COVID-19 symptoms | 8 months
  COVID-19 symptoms assessed through binary questions, asking presence or not of fever (≥ 38 Celsius), cough, shortness of breath and other symptoms.
  For both phases.
Psychological stress | 8 months
  Psychological stress is assessed using a verbal anxiety scale (EVA in French) ranging from 0 (no anxiety) to 10 (severe anxiety).
  For both phases.
Social Isolation | 8 months
  Social isolation is assessed through accessibility to medication, food and home care.
  For both phases.
Caregiver burden | 8 months
  Caregiver burden using the 4-item scale of the Caregiver Burden Interview.
  For both phases.
Number of completed questionnaires and recommendations given | 8 months
  By summing up the number of completed questionnaires and recommendations given.
  For both phases.
Number of recommendations followed by participants | 8 months
  By summing up the number of recommendations followed by participants.
  For both phases.
Loss of autonomy | 8 months
  The level of loss of autonomy is assessed by two scales :
  * Activities of Daily Living (ADL) scale score from 0 (very dependent) to 6 (very independent)
  * Instrumental Activities of Daily Living (IADL) scale score from 0 (not autonomous) to 4 (autonomous)
  For both phases.
Quality of life of participants | 8 months
  Quality of life is assessed by EuroQol-5D (EQ-5D), a standardized measure of health developped by EuroQol group. EQ-5D is composed of two parts :
  * a short survey with 5 questions giving a score from 1 (no problem) to 5 (severe problem)
  * a visual scale that ranges from 0 (worst health that participant can ever imagine) to 100 (best health participant can ever imagine).
  For both phases.
Consumption of services and care resources | 8 months
  Consumption of services and care resources measured by :
  * the intervention (number and type) in the participant home of one or more community organizations
  * the number and type of consultations made with a professional (doctor, nurse, physiotherapist, etc.) reported by the caregiver
  * the number of visits to the emergency department and the number of hospitalizations reported by the caregiver.
  For both phases.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No